CLINICAL TRIAL: NCT06247137
Title: Evaluation of the Effect of a Food Supplementation With a Combined Food Supplement on Lipid Pattern, Indexes of Non-alcoholic Fatty Liver Disease and Systemic Inflammation in Healthy Subjects With Suboptimal LDL-C Levels: a Two-arm Double-blind, Placebo- Controlled, Randomized, Clinical Trial
Brief Title: Effect of a Food Supplementation With a Combined Food Supplement on Lipid Pattern, Indexes of Non-alcoholic Fatty Liver Disease and Systemic Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Claudio Borghi, Prof. Dr., University of Bologna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NUT1-BO-2021
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dietary supplement (Active Comparator)
  Interventions: Dietary Supplement: Dietary Supplement
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary Supplement — Dietary supplement formulated with components of natural origin: artichoke, bergamot, folic acid, astaxanthin, Chromium picolinate and excipients.
  Oral administration: 1 tablet/day at evening meal
  Arms: Dietary supplement
Other: Placebo — Placebo (microcrystalline cellulose, calcium carbonate, magnesium stearate, silica dioxide and iron oxides).
  Oral administration: 1 tablet/day at evening meal.
  Arms: Placebo

SUMMARY:
Several controlled interventional studies have shown that there is a close correlation between cholesterol reduction and cardiovascular risk; in fact, reductions in serum levels of total cholesterol and low-density lipoprotein cholesterol (LDL-C), obtained through lifestyle modification or specific drugs, result in reductions in the incidence of major coronary events. The effectiveness of these interventions has been demonstrated both in subjects in primary prevention and in subjects in secondary prevention.

Based on this evidence, the National Cholesterol Education Program (NCEP) has defined in the ATP III report the target values of LDL-C to be reached with interventions on food and / or pharmacological habits to perform an effective cardiovascular prevention.

Although the atherogenic action of hypercholesterolemia is largely attributable to a direct damage exerted on vascular endothelium, recent studies suggest that the activation of a low-grade systemic pro-inflammatory state, typical of the patient with cardiovascular risk factors, does also play a role in the determinism of endothelial damage and atheroma degeneration of the arteries. It is believed that this systemic inflammation, as documented by the determination of some humoral signs of inflammation (e.g. C-reactive protein, interleukin-6, tumor necrosis factor-α), may further contribute to an increase of cardiovascular risk.

The inflammatory state can modulate the atherosclerotic process at various levels, determining endothelial activation, promoting leukocyte chemotaxis in the sub-intimal space of the arterial wall and therefore the formation of an atheromatous plaque rich in inflammatory cells; the latter represents the lesion responsible for the vast majority of the coronary and cerebrovascular events observed in subjects with cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects agree to participate in the study and having dated and signed the informed consent form.
2. Subjects who have the capability to communicate, to make themselves understood, and to comply with the study's requirements.
3. Male or female aged ≥ 18 years and ≤ 70 years old.
4. LDL-Cholesterol blood levels >115 mg/dL and < 190 mg/dL.
5. TG<400 mg/dL.
6. Subjects who, according to the SCORE charts, have a low or moderate cardiovascular risk (defined as a total cardiovascular risk < 5%) and for whom, according to ESC/EAS guidelines 2012, the intervention strategy does not require a pharmacological lipid-lowering intervention.
7. Patient covered by the Social Security scheme.

Exclusion Criteria:

1. Subjects already affected by cardiovascular diseases (secondary prevention) or with estimated 10 years cardiovascular disease risk> 5%;
2. Obesity (BMI>30 kg/m2) or diabetes mellitus;
3. Assumption of lipid lowering drugs or food supplements, or drugs potentially affecting the lipid metabolism;
4. Antihypertensive treatment not stabilized since at least 3 months;
5. Anticoagulants therapy
6. Uncontrolled hypertension (systolic blood pressure> 190 mmHg or diastolic arterial pressure> 100 mmHg);
7. Known current thyroid, gastrointestinal or hepatobiliary diseases;
8. Any medical or surgical condition that would limit the patient adhesion to the study protocol;
9. Abuse of alcohol or drugs (current or previous);
10. History of malignant neoplasia in the 5 years prior to enrolment in the study;
11. History or clinical evidence of inflammatory disease such as severe arthritis, systemic lupus erythematosus or chronic inflammatory diseases or current therapy with immunosuppressive agents or long-term glucocorticoids;
12. History or clinical evidence of any significant concomitant disease that could compromise the safety of the subject or the possibility of completing the study;
13. Known previous intolerance to one component of the tested nutraceuticals
14. Women in fertile age not using consolidated contraceptive methods
15. Pregnancy and Breastfeeding.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
LDL-cholesterolemia reduction from baseline and between groups | 3 months
  Reduction of LDL-cholesterolemia after 3 months of treatment

SECONDARY OUTCOMES:
LDL-cholesterolemia reduction from baseline and between groups at 6 weeks | 6 weeks
  Reduction of LDL-cholesterolemia after 6 weeks of treatment
Changes in hsCRP | 3 months
  Evaluate the effect of the dietary supplementation on blood levels of hsCRP after 3 months of treatment
Change in vascular reactivity | 3 months
  Evaluate the effect of the dietray supplementation on the vascular reactivity (Endocheck®)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Borghi, MD, Principal Investigator — University of Bologna
Locations (1):
- University of Bologna, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: No